CLINICAL TRIAL: NCT03528291
Title: Decision Relevance of Transient Circulatory Support for Acute Cardiogenic Shock: Patients' Characteristics and Follow-up
Brief Title: Transient Circulatory Support in Cardiogenic Shock
Acronym: ALLOASSIST
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: 9842
Record Dates: First submitted 2018-02-19; First posted 2018-05-17 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Acute Cardiogenic Shock
Keywords: Human,; adult,; intensive care unit,; cardiogenic shock,; Transient circulatory support,; extra corporeal life support; Impella
MeSH Terms: conditions — Shock, Cardiogenic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cardiogenic shock treated with medical treatment: Patients with cardiogenic shock treated only by medical treatment
- Cardiogenic shock treated with transient circulatory support: Patients where transient circulatory support was implanted: veno-arterial extracorporeal circulatory life support (ECLS), Impella

SUMMARY:
The purpose of this multicenter prospective study is to determine if the decision of transient circulatory support (TCS) in cardiogenic shock is relevant. TCS is a recommended treatment of refractory cardiogenic shock but precise indications are not definitively founded. Some studies described patients with TCS in order to establish mortality predictive scores (ENCOURAGE, SAVE), but no study has assessed the clinical relevance of the TCS decision yet. Therefore, The investigators propose to compare the characteristics and the follow-up of patients in acute cardiogenic shock, once TCS implantation was decided or not by the heart team.

DETAILED DESCRIPTION:
This French multicenter prospective observational study is aimed at determining if the decision of transient circulatory support (TCS) in cardiogenic shock is pertinent, i.e. at least as effective as the medical treatment.

All patients with cardiogenic shock for whom indication of TCS was discussed within the multidisciplinary heart team (cardiologist, intensivist and cardiac surgeon) are consecutively included in the study.

Two groups of patients are defined:

* Patients with cardiogenic shock treated by medical treatement
* Patients with cardiogenic shock treated by TCS (extracorporeal circulatory life support and/or Impella).

The main objective is to compare mortality between the 2 groups. Secondary objectives are ICU follow-up characteristics and quality of life questionnaire at day 180.

Statistical analysis will include a propensity-matched method to compare the groups to avoid confounding factors. The number of necessary subjects (n=240, 120 in each group) was calculated assuming that TCS has a superiority of 20% in comparison with medical treatment in severe cardiogenic shock, with a study power of 80%, and an alpha risk of 5%.

ELIGIBILITY:
Inclusion Criteria:

* Cardiogenic shock :

  • Systolic BP<90mmHg despite adequate filling pressure
* Or need of cathecolamines to maintain SBP > 90mmHg

  * Signs of right-sided and/or left-sided congestion
  * Signs of tissue hypoperfusion : oliguria, cold sweated extremities, mental confusion, dizziness, narrow pulse pressure, blood lactate > 2 mmol/L
* Short-term mechanical circulatory support discussed by the multidisciplinary heart team

Exclusion Criteria:

* Post cardiotomy cardiogenic shock
* Refractory cardiac arrest
* Cardiac Arrest with No Flow >3 min and/or non shokable rythm
* Contraindication to transient circulatory support because of comorbidities, neurological dysfunction, severe end-organ failure or aortic regurgitation
* Pregnant or brest-feeding women,
* Age < 18 year-old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in cardiogenic shock for whom transient circulatory support was discussed within the multidisciplinary heart team
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2017-07-12 (Actual); Primary Completion 2021-10-31 (Estimated); Study Completion 2021-10-31 (Estimated)

PRIMARY OUTCOMES:
Hospital Mortality | From inclusion day to day 180
  Mortality rate in the 2 groups at the time of hospital discharge

SECONDARY OUTCOMES:
Short term mortality rate | From inclusion day to Intensive Care Unit (ICU) discharge or day 28 whichever came first
  Mortality rate at day 28
Acute renal failure | From inclusion day to ICU discharge or day 28 whichever came first
  Incidence of renal replacement therapy
Respiratory failure | From inclusion day to ICU discharge or day 28 whichever came first
  Days of mechanical ventilation
Thromboembolic events | From inclusion day to ICU discharge or day 28 whichever came first
  Incidence of stroke, peripheral or mesenteric ischemia
Bleeding events | From inclusion day to ICU discharge or day 28 whichever came first
  Incidence of red blood cell transfusion
ICU stays | From inclusion day to day 180
  Length of stay in ICU (number of days)
Hospital stays | From inclusion day to day 180
  Length of stay in hospital (number of days)
Quality of life score SF 36 | From inclusion day to day 180
  Quality of life, evaluated by the Short Form Survey scoring (SF36 score) using the RAND 36-Item Health Survey 1.0, which will be sent by mail at day 180 after inclusion.
  The RAND 36-Item Health Survey (Version 1.0) taps eight health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. It also includes a single item that provides an indication of perceived change in health. Each item is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100, respectively.
Long term mortality rate | From inclusion day to day 180
  Mortality rate at day 180

CONTACTS AND LOCATIONS:
Overall Officials: Jacob ELIET, M.D, Principal Investigator — Montpellier Academic Hospital Department of Anesthesia-Resuscitation Arnaud de Villeneuve
Locations (1):
- Department of Anesthesia-Resuscitation Arnaud de Villeneuve, Montpellier, France

REFERENCES:
- [Derived] Ughetto A, Eliet J, Nagot N, David H, Bazalgette F, Marin G, Kollen S, Mourad M, Zeroual N, Muller L, Gaudard P, Colson P. Early temporary mechanical circulatory support for cardiogenic shock: Real-life data from a regional cardiac assistance network. J Heart Lung Transplant. 2024 Jun;43(6):911-919. doi: 10.1016/j.healun.2024.02.009. Epub 2024 Feb 15. PMID 38367739